CLINICAL TRIAL: NCT02900131
Title: Efficacy, Safety and Dose Finding Trial of Topical Jaungo Application in Atopic Dermatitis Patients: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy, Safety and Dose Finding Trial of Topical Jaungo Application in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, In-Hwa Choi, Clinical Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISEE_2015_JWG
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — jaungo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- trial group 1 (Experimental): Participants will receive Jaungo and placebo once a day for three weeks.
  Interventions: Drug: Jaungo; Drug: Placebo
- trial group 2 (Experimental): Participants will receive Jaungo twice a day for three weeks.
  Interventions: Drug: Jaungo
- control group (Placebo Comparator): Participants will receive placebo twice a day for three weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaungo — Participants in trial group 1 will apply Jaungo and placebo to the lesion once a day for three weeks. Participants in trial group 2 will apply Jaungo to the lesion twice a day for three weeks.
  Other Names: Hanpoong Jaungo
  Arms: trial group 1; trial group 2
Drug: Placebo — Participants in trial group 1 will apply Jaungo and placebo to the lesion once a day for three weeks. Participants in control group will apply placebo to the lesion twice a day for three weeks.
  Other Names: Jaungo placebo
  Arms: control group; trial group 1

SUMMARY:
Atopic Dermatitis is a chronic relapsing eczematous skin disease with increasing prevalence. Complementary and alternative medical approaches have been employed to relieve symptoms of Atopic Dermatitis. We aim to establish basic clinical efficacy and safety data for Jaungo in patients with Atopic Dermatitis.

DETAILED DESCRIPTION:
This study is a randomised, double blind, placebo-controlled, single-centre trial with three parallel arms (trial group 1, trial group 2, and control group). The diagnosis of Atopic Dermatitis will be made according to the criteria of Hanifin and Rajka. Participants will receive Jaungo or a placebo-drug for three weeks. Participants in trial group 1 will apply Jaungo and placebo to the lesion once a day for three weeks. Participants in trial group 2 will apply Jaungo to the lesion twice a day for three weeks. Participants in control group will apply placebo to the lesion twice a day for three weeks. Each participant will be examined for EASI (Eczema area and severity index), SCORAD (SCORing of Atopic Dermatitis), TEWL (Transepidermal water loss) and DLQI (Dermatology Life Quality Index) before and after applying medication. The outcomes to evaluate the maintenance of safety are Draize score, blood test and expert's opinion.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of AD will be made according to the criteria of Hanifin and Rajka
2. Age: 5 years to 65 years
3. objective SCORAD ≦40, Diagnosis of Mild to Moderate Atopic Dermatitis (AD)
4. Exoriation≥1, Lichenification≥1, Dryness≥1 or Exoriation+Lichenification+Dryness≥3
5. Participants who able to express intention
6. Participants willing to provide written informed consent

Exclusion Criteria:

1. Participants have oozing in the lesion
2. Users of following medications prior to trial periods

   ① Oral steroids, immunosuppressants and antibiotics within 4 weeks prior to this trial

   ② Topical steroids, immunosuppressants and antibiotics within 2 weeks prior to this trial

   ③ Light therapy within 2 weeks prior to this trial

   ④ Other medications thought to be inappropriate by researchers
3. Participants have severe burn or wide wound
4. Participants have oozing or ulcer in the lesion
5. Allergic reactions to Angelica gigas, Siebold et Zuccarini, sesame oil and lard
6. Participants have skin disease except atopic dermatitis
7. Participants have severe renal function disease (sCr > 2.0 mg/dL)
8. Participants have severe liver function disease (ALT, AST, ALP ≥ 2.5 × normal limits)
9. Participants have uncontrolled chronic diseases
10. Pregnancy, lactation
11. Participation in another clinical trial within one month of enrolment
12. Underlying disease or history of severe disease, abnormal state (paralysis; mental retardation other emotional or mental problems; diseases that can affect the absorption of drugs; no enough time to participate in this trial; visual disturbance and hearing impairment; inability to understand written consent or engage in this study)
13. Judgment by experts that the potential subject's participation is inappropriate.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 'Eczema area and severity index (EASI)' | Visit2(scheduled within a week of baseline), Visit3(in 3 weeks after visit2)

SECONDARY OUTCOMES:
Change from baseline in 'SCORing of Atopic Dermatitis (SCORAD)' | Visit2(scheduled within a week of baseline), Visit3(in 3 weeks after visit2)
Change from baseline in 'Transepidermal water loss (TEWL)' | Visit2(scheduled within a week of baseline), Visit3(in 3 weeks after visit2)
Change from baseline in 'Dermatology Life Quality Index (DLQI)' | Visit2(scheduled within a week of baseline), Visit3(in 3 weeks after visit2)
Change from baseline in 'Total IgE' | Visit1, Visit3(in 3 weeks after visit2)
The clinical phenotype evaluation system of atopic dermatitis | Visit2(scheduled within a week of baseline)
  Evaluation based on the results of 'clinical phenotype evaluation system of atopic dermatitis' questionnaire
Change from baseline in 'eosinophil count' | Visit1, Visit3(in 3 weeks after visit2)
Change from baseline in 'IL-17' | Visit1, Visit3(in 3 weeks after visit2)
Change from baseline in 'IL-22' | Visit1, Visit3(in 3 weeks after visit2)
Change from baseline in 'IFN-γ' | Visit1, Visit3(in 3 weeks after visit2)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Kyu Ko, KMD, PhD, Study Chair — Kyunghee University
Locations (1):
- Kyung Hee University Hospital, Seoul, Hoegi, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yun Y, Ko Y, Ahn JH, Jang BH, Kim K, Ko SG, Choi I. Topical application of Jaungo in atopic dermatitis patients: study protocol for a randomized, controlled trial. Trials. 2017 Apr 12;18(1):176. doi: 10.1186/s13063-017-1920-9. PMID 28403910